CLINICAL TRIAL: NCT05023239
Title: The Effect of Ultrasound-Guided Suprazygomatic Maxillary Nerve Block for Minimize the Post-operative Pain in Tonsillectomy Surgery
Brief Title: Ultrasound-Guided Suprazygomatic Maxillary Nerve Block as A Part of Multimodal Analgesic Regimens
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Amr Samir Wahdan, Lecturer of Anesthesia, Pain management and Surgical ICU, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: n-2021
Record Dates: First submitted 2021-08-21; First posted 2021-08-26 (Actual); Last update posted 2021-08-26 (Actual); Status verified 2021-08

CONDITIONS: Suprazygomatic Maxillary Nerve Block

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Sham Comparator): patients will receive sham block by 10 ml of normal saline (5 mL in each side) as a control.
  Interventions: Other: UG-SZM Group
- UG-SZM Group (Experimental): The patients will be receive bilateral Ultrasound-Guided Suprazygomatic Maxillary (UG-SZM) Nerve Blocks 10 mL of a local anesthetic mixture composed of 0.25% plain bupivacaine
  Interventions: Other: UG-SZM Group

INTERVENTIONS:
Other: UG-SZM Group — The patients will be receive Ultrasound-Guided Suprazygomatic Maxillary Nerve Blocks 10 mL of a local anesthetic mixture composed of 0.25% plain bupivacaine .

SUMMARY:
Inadequate peri-operative analgesia may contribute to an increased risk of bleeding, suture dehiscence and unacceptable surgical outcomes. Moreover, these patients are at high risk of postoperative airway obstruction and respiratory failure.

Opioids may contribute to these complications. Appropriate use of regional anaesthesia may mitigate or eliminate many of these concerns. The maxillary nerve is responsible for the sensory innervation of the midface, including the hard and soft palates, upper jaw, upper dental arch and upper lip.Recently, the successful use of maxillary nerve block by the suprazygomatic approach has been reported in children undergoing cleft palate surgery. However, the use of this block has not been described in large series of patients, and the effectiveness of the suprazygomatic approach has not been evaluated in patients undergoing tonsillectomy .

ELIGIBILITY:
* Inclusion criteria

  1. Pediatric patients aged 4-12 years
  2. Genders eligible for study: both sexes
  3. ASA physical status I and II
  4. Undergoing tonsillectomy surgery

     Exclusion criteria
* Parents' refusal
* Contraindications to regional anesthesia
* Known allergy to local anesthetics
* Bleeding disorders
* Children with diabetes mellitus, obstructive sleep apnea syndrome, cardiac, renal, liver or blood diseases, swallowing disorders or peritonsillar abscess,
* Children receiving regular analgesia within the last week before surgery,
* Children undergoing simultaneous procedure in the field of surgery like adenoidectomy or tongue tie will be all excluded from the study.

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 52 (Estimated)
Dates: Start 2021-10-01 (Estimated); Primary Completion 2022-10-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
postoperative Meperidine consumption | 24 hours
  total dose of Meperidine consumption

SECONDARY OUTCOMES:
incidence of complication | 24 hours
  postoperative complication

IPD SHARING:
Plan to Share IPD: Undecided